CLINICAL TRIAL: NCT07247279
Title: A Multicenter Non Interventional Single Arm Retrospective-prospective Observational Study in Therapeutic Approaches in AChR-Antibody Positive Generalized Myasthenia Gravis (gMG) in Real Clinical Practice in Russia
Brief Title: Epidemiological Study of Treatment Approaches in AChR-Antibody Positive Generalized Myasthenia Gravis in Russia
Status: Recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D9281R00003
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Rare Diseases; Generalized Myasthenia Gravis (gMG)
MeSH Terms: conditions — Rare Diseases; Myasthenia Gravis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

SUMMARY:
This is a multicenter, non-interventional, retrospective-prospective, single-arm observational study designed to describe real-world treatment approaches and clinical outcomes among adults with acetylcholine receptor (AChR) antibody-positive generalized myasthenia gravis (gMG) in routine clinical practice in Russia.

DETAILED DESCRIPTION:
This is a multicenter, non-interventional, retrospective-prospective, single-arm observational study designed to describe real-world treatment approaches and clinical outcomes among adults with acetylcholine receptor (AChR) antibody-positive generalized myasthenia gravis (gMG) in routine clinical practice in Russia.

The primary objective is to characterize the demographic and clinical profile of adult AChR-Ab-positive gMG patients. Key secondary objectives include assessing disease severity over time (MG-ADL, QMG, MGFA class), evaluating rates, duration, and reasons for all-cause and gMG-related hospitalizations, describing diagnostic pathways and treatment strategies (including first-line regimens and use of therapies such as anticholinesterase agents, corticosteroids, immunosuppressants, IVIG, plasmapheresis/plasma filtration, thymectomy, rituximab, and complement C5 inhibitors), exploring patterns and outcomes of myasthenic crises, and documenting meningococcal vaccination and any prophylactic antibiotic use prior to initiation of C5 inhibitor therapy.

Approximately 100 adults will be enrolled consecutively across about 10 specialized sites. The study will sequentially include only those patients who have signed the informed consent form (ICF). Eligible patients will be enrolled consecutively at each site to minimize selection bias. Data are collected from existing paper/electronic medical records (secondary data collection) and recorded into an eCRF at seven timepoints: baseline (with retrospective abstraction, including medical history from diagnosis) and prospective follow-up every 6 months up to Month 36 (±1 month windows). No study-mandated interventions, tests, or visit schedules are imposed; all care follows routine practice.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥18 years) diagnosed with generalized MG positive for acetylcholine receptor (AChR) antibodies.
2. Provision of signed and dated written informed consent.

Exclusion Criteria:

1. Participants currently enrolled in clinical studies for treatment of gMG.
2. Ocular MG only.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants of both sexes aged 18 years and older with diagnosis of AChR-antibody positive generalized MG will be enrolled in various clinical institutions in Russia that provide treatment for gMG patients.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2025-12-23 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Age at baseline (years) | Baseline (Month 0; at informed consent and enrollment)
  Patient age in full years at study enrollment (ICF signing). Summarized as a quantitative variable and as categorical distribution by ≤50 years vs >50 years.
Age at gMG diagnosis (years) | Baseline (retrospective abstraction at Month 0)
  Patient age in full years at the date of generalized myasthenia gravis (gMG) diagnosis. Summarized as a quantitative variable and as categorical distribution by ≤50 years vs >50 years.
Sex and ethnicity distribution | Baseline (Month 0)
  Proportion of patients by sex (male, female) and ethnicity (White, Asian, Black, other) recorded at enrollment.
Body Mass Index (BMI) | Baseline (Month 0; last available measurements closest to ICF signing)
  BMI in kg/m^2 calculated as weight (kg)/height (m)^2 using the most recent values closest to enrollment, summarized as mean, SD, median, IQR, minimum, maximum. Height and weight are abstracted from medical records.
Disease duration (days) | Baseline (Month 0)
  Time between the date of documented gMG diagnosis and the date of informed consent/enrollment, summarized as median and IQR (and mean, SD, min, max). Calculated in months/years based on dates abstracted from medical records to the eCRF.
Clinical symptom profile of gMG | Baseline (Month 0)
  Proportion of patients presenting each predefined gMG symptom category at enrollment (ocular, bulbar, respiratory, chewing/facial, limb/trunk/neck weakness, autonomic dysfunction subdomains); summarized as counts and percentages.
Comorbidity profile | Baseline (Month 0)
  Proportion of patients with specified comorbidities in history or present at enrollment: autoimmune thyroiditis/hyperthyroidism, systemic lupus erythematosus, rheumatoid arthritis, autoimmune encephalitis, arterial hypertension, hyperlipidemia.
Number and proportion of patients with gMG-related hospitalizations | Retrospective period from gMG diagnosis to Baseline (Month 0)
  Patients with ≥1 hospitalization attributed to gMG (investigator judgment) from date of gMG diagnosis to ICF signing.
Duration of gMG-related hospitalizations (days) | Retrospective period from gMG diagnosis to Baseline (Month 0)
  Sum of days of gMG-related hospitalizations per patient from gMG diagnosis to ICF signing.

SECONDARY OUTCOMES:
MG-ADL total score and change from baseline | Baseline (Month 0) and Months 6, 12, 18, 24, 30, 36 (±1 month)
  Patient-reported MG-ADL total score (range 0-24; higher=worse). Report descriptive statistics at each time point and change from Baseline (visit value minus Baseline). Scores are abstracted from routine care records; only total scores documented in source are collected.
QMG total score and change from baseline | Baseline (Month 0) and Months 6, 12, 18, 24, 30, 36 (±1 month)
  Physician-reported QMG total score (0-39; higher=worse). Metrics: absolute score and change from baseline. Summarized descriptively. Collected only if present in routine practice records.
Distribution of MGFA clinical classification over time | Baseline (Month 0) and Months 6, 12, 18, 24, 30, 36 (±1 month)
  Proportion of participants in each MGFA class (I, IIa/IIb, IIIa/IIIb, IVa/IVb, V) at each time point. Also report proportion improving (lower class) or worsening (higher class) versus Baseline. MGFA class is abstracted only if recorded in routine practice.
Number and proportion of patients with all-cause hospitalization | From Baseline through Months 6, 12, 18, 24, 30, 36 (±1 month)
  Patients experiencing ≥1 hospitalization for any cause during prospective follow-up. Metric: count and proportion (percentage) of patients with ≥1 event. Each participant's status (yes/no) assessed across the follow-up period.
Duration of all-cause hospitalizations (days per participant) | From Baseline through Months 6, 12, 18, 24, 30, 36 (±1 month)
  Total days hospitalized for any cause per participant during prospective follow-up. Metric: sum of hospital-day durations per participant; summarized descriptively.
Number and proportion of patients with gMG-related hospitalization | From Baseline through Months 6, 12, 18, 24, 30, 36 (±1 month)
  Patients with ≥1 hospitalization attributed to gMG during follow-up. Categorize reasons: related to MG exacerbation (myasthenic crisis) vs not related (thymectomy, investigation, social reason, other). Record ICU admission for gMG-related hospitalizations (yes/no). Report count and proportion (percentage) of affected patients overall and by categories.
Duration of gMG-related hospitalizations (days per participant) | From Baseline through Months 6, 12, 18, 24, 30, 36 (±1 month)
  Total days hospitalized for gMG-related reasons per participant during prospective follow-up. Metric: sum of hospital-day durations for gMG-related stays; summarized descriptively.
Time from MG symptom onset to gMG diagnosis (months) | Retrospective period prior to Baseline
  Interval between the date of first MG symptoms/suspicion (if known) and the date of generalized MG (gMG) diagnosis. Metric: duration in months (or days if available); summarized descriptively. Evaluated only for patients with a documented onset date.
Prior misdiagnoses before gMG diagnosis (number and proportion by category) | Retrospective period prior to Baseline
  Proportion of participants with ≥1 prior misdiagnosis and distribution by category (myopathies, polyneuropathies, Lambert-Eaton, mitochondrial encephalomyopathies, congenital myasthenic syndromes, cerebrovascular accidents, brainstem encephalitis, brain tumors, ALS).
Diagnostic examinations for gMG confirmation and available results | Retrospective period prior to Baseline
  Proportion with each examination and latest available result: AChR-Ab (required positive), CT/MRI chest/mediastinum, brain/spinal MRI, ENMG, single-fiber EMG, RNS. Report counts, percentages (95% CI), and result categories if available.
Diagnostic test usage and results | Retrospective period prior to Baseline
  Proportion with each test performed and latest result (positive/negative/unknown) as documented in routine care; report counts and percentages with 95% CI.
Drug therapies received (proportion by class) | 12 months pre-Baseline and Baseline to Month 36 (±1 month)
  Proportion of patients receiving each therapy class: anticholinesterase (neostigmine), IVIG, corticosteroids (prednisolone/methylprednisolone), complement inhibitors (ravulizumab/eculizumab), diuretics, potassium, immunosuppressants (e.g., azathioprine, mycophenolate, cyclosporine), rituximab. Summarized as counts/percentages by class.
Duration of drug therapies (days per participant) | 12 months pre-Baseline and Baseline to Month 36 (±1 month)
  For each therapy class received, total days on therapy per participant during the assessment window; summarized descriptively.
Mean daily corticosteroid dose (prednisolone equivalent) | 12 months pre-Baseline and Baseline to Month 36 (±1 month)
  Among CS users, average daily dose recorded in mg; convert methylprednisolone to prednisolone equivalent for analysis. Summarized with descriptive statistics.
Plasmapheresis/plasma exchange/plasmafiltration use (proportion) | 12 months pre-Baseline and Baseline to Month 36. (±1 month)
  Proportion of patients receiving plasmapheresis, plasma exchange, or plasmafiltration for gMG; summarized as counts and percentages.
Duration of plasmapheresis/plasma exchange/plasmafiltration (days) | 12 months pre-Baseline and Baseline to Month 36 (±1 month)
  Total treatment days per participant for plasmapheresis, plasma exchange, or plasmafiltration within the assessment window; summarized descriptively.
Thymectomy performed | 12 months pre-Baseline and Baseline to Month 36 (±1 month)
  Proportion of patients who underwent thymectomy for gMG; summarized as counts and percentages.
Invasive lung ventilation required | 12 months pre-Baseline and Baseline to Month 36 (±1 month)
  Proportion of patients requiring invasive mechanical ventilation for gMG; summarized as counts and percentages.
First-line treatment regimen at gMG diagnosis | At gMG diagnosis (retrospective abstraction at Baseline)
  Distribution of initial treatment components at diagnosis (same therapy categories as above); summarized as counts and percentages by regimen.
Myasthenic crisis in prior 12 months | 12 months prior to Baseline (Month 0)
  Proportion with ≥1 crisis and distribution by number of episodes (1, 2, ≥3) during the 12 months prior to enrollment; counts and percentages from medical records.
Myasthenic crisis during follow-up | From Baseline to Month 36 (±1 month)
  Proportion with ≥1 crisis and distribution by number of episodes (1, 2, ≥3) during prospective follow-up; counts and percentages from medical records.
Crisis precipitants-physical stressors | 12 months pre-Baseline and Baseline to Month 36 (±1 month)
  Proportion of crisis episodes associated with predefined physical precipitants: aspiration pneumonitis, infection, perimenstrual state, pregnancy, sleep deprivation, surgery, environmental stressors, emotional stress, pain, temperature extremes, tapering of immune-modulating medications.
Crisis precipitants-medications | 12 months pre-Baseline and Baseline to Month 36 (±1 month)
  Proportion of crisis episodes associated with predefined medications: α-interferon; antibiotics (e.g., aminoglycosides, macrolides, quinolones, polymyxin); antiepileptics (e.g., gabapentin, phenytoin, carbamazepine, high-dose benzodiazepines); β-blockers; calcium channel antagonists; contrast media; magnesium; hormonal drugs (e.g., corticosteroids, ACTH, oral contraceptives, oxytocin, thyroid hormones); antithyroid agents; antiarrhythmics (e.g., procainamide, quinidine).
Crisis outcomes by MGFA class change | Months 6, 12, 18, 24, 30, 36 (±1 month)
  Change in MGFA class from the most recent pre-crisis assessment to the nearest post-crisis scheduled assessment; proportion improved, unchanged, or worsened.
Initiation of complement C5 inhibitor therapy (C5IT) | From gMG diagnosis to Month 36 (±1 month)
  Proportion of participants who initiated C5IT during observation; counts and percentages; with start/stop dates abstracted from records.
Meningococcal vaccination prior to C5IT initiation | From gMG diagnosis to C5IT start (vaccination events abstracted during follow-up)
  Among those who initiated C5IT, proportion with documented meningococcal vaccination before first dose; time from gMG diagnosis to first vaccination; record revaccinations. Report counts, percentages, and time-to-vaccination summary.
Prophylactic antibiotic use prior to C5IT initiation | From gMG diagnosis to C5IT start (antibiotic events abstracted during follow-up)
  Among those who initiated C5IT, proportion with documented prophylactic antibiotic use prior to first dose; time from gMG diagnosis to first prophylactic use; record repeated prophylaxis. Report counts, percentages, and time-to-prophylaxis summary.

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - Research Site, Kazan'
  - Research Site, Novosibirsk

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/